CLINICAL TRIAL: NCT01284270
Title: High Amount of Lipid Rich Necrotic Core Lesion Identified by Pre-interventional Intravascular Ultrasound (IVUS) is Associated With High Rate of Delayed Hyper-enhancement as Detected by Contrast-enhanced Cardiac Magnetic Resonance Imaging
Brief Title: Lipid Rich Necrotic Core Lesion Detected by Cardiac Magnetic Resonance Imaging (CMR)
Acronym: Hawaii
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not to be initiated
Sponsor: Piedmont Healthcare (Other)
Collaborators: Volcano Corporation (Industry); GE Healthcare (Industry); Siemens Medical Solutions (Industry)
Responsible Party: Szilard Voros, MD, Piedmont Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Hawaii
Record Dates: First submitted 2011-01-21; First posted 2011-01-26 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2011-06

CONDITIONS: Coronary Disease
Keywords: Cardiac MRI; Plaque
MeSH Terms: conditions — Coronary Disease; Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Patients (Other): All patients undergo the same study procedures
  Interventions: Other: Cardiac MRI

INTERVENTIONS:
Other: Cardiac MRI — Cardiac MRI

SUMMARY:
The purpose of this study is to evaluate whether some features of plaques in coronary arteries predispose the heart muscle to injuries during angioplasty in patients with a narrowing in at least one of the arteries that may need a stent placed during a heart catheterization. Participants undergo a cardiovascular magnetic resonance imaging (MRI) study before the heart catheterization to look for scarring in the heart muscle. During the heart catheterization, participants undergo an intravascular ultrasound (IVUS) exam to look at the make-up of the plaques before the stent placement and the investigators will measure the pressures in the arteries to look at how severe the blockage is. Within 30 days after the heart catheterization, participants will have a second MRI done to look for any new scar in the heart muscle.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 90 years
* Patients with known obstrucive coronary arterial disease for PCI in a native coronary artery
* Ability and willingness to consent and Authorization for use of personal health information (PHI)
* Ability and willingness to the required follow up procedures

Exclusion Criteria:

* An acute myocardial infarction in the vascular territory of interest.
* History of percutaneous coronary intervention in the major epicardial vessel of interest
* Lesion characteristics that preclude IVUS
* The presence of delayed enhancement in the territory of the study vessel on baseline CMR
* Patients with current history of cardiomyopathy which is known to cause enhancement on CMR study
* Patients who are considered hemodynamically unstable based on clinical assessment by the physician
* Patients with Class IV congestive heart failure at time of enrollment
* Patients with poorly controlled hypertension with SBP >/= 210mmhg and/or DBP >/=140 hypertension unable to be treated, at time of enrollment
* GFR</=30 pre-procedure per institutional standards
* Patients with any known co-morbid conditions that is limiting their life expectancy to < 1year
* A known contraindication to Adenosine, including but not limited to:
* Moderate to severe hyperactive airway disease such as asthma and severe COPD
* Second or third degree AV block
* Known sinus node disease, such as sick sinus syndrome or symptomatic bradycardia
* Known hypersensitivity to Adenosine
* A known contraindication to MRI
* Electronically, magnetically, and mechanically activated implants
* Ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators, and cardiac pacemakers
* Metallic splinters/fragments in sensitive tissues including the eye, brain, spinal cord etc…
* Ferromagnetic haemostatic clips in the central nervous system
* A known contraindication to Gadolinium
* Patients with history of allergic reactions to gadolinium based contrast
* Patients with glomerular filtration rate (GFR) </= 30ml/min
* Inability or unwillingness to consent and Authorization for use of PHI
* Patients who are unwilling or unable to follow up
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the occurrence of new areas of infarction (heart attack) in the heart muscle supplied by the vessel that was treated. | 6 months

SECONDARY OUTCOMES:
Evaluate the occurrence of new areas of infarction (heart attack) in the heart muscle supplied by any of the 3 major blood vessels of the heart | 6 months